CLINICAL TRIAL: NCT00800813
Title: Assessing the Change in Penile Length Following Bilateral Nerve-Sparing Radical Prostatectomy
Brief Title: Change in Penile Length Following Bilateral Nerve-Sparing Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-135
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; Erectile function; Peyronie's Plaque; 08-135
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- open, laparoscopic, or robotic-assisted lap: Patients will also be assessed for penile length and the presence of Peyronie's Disease at these specified times.
  Interventions: Behavioral: Penile Exam, Peyronie's Plaque and Erectile function assessment

INTERVENTIONS:
Behavioral: Penile Exam, Peyronie's Plaque and Erectile function assessment — At the baseline visit, the patient's co-morbidities, height, weight with calculation of body mass index will be documented.
  After surgery, the patient will be instructed to keep a diary to record erectile function including how often they use a PDE-5 inhibitor or injection therapy and each time they get an erection and the level of rigidity. The diary is required to document PDE-5 inhibitor and injection therapy use and response in each sexual encounter, unlike the IIEF questionnaire, which addresses erectile function over a 4-week period. Accurate documentation is essential for erectile function assessment, as patient choice of erectile function medication may differ in each sexual encounter, and accordingly, the achieved rigidity level.

SUMMARY:
Some men complain of changes in the shape or dimensions of their penis after undergoing radical prostatectomy (removal of the prostate) for prostate cancer. Changes in penile dimensions include shortening or decreased girth. Changes in shape include a curvature or bending of the penis, and/or the appearance of indentation. These changes may be associated with formation of scar tissue involving the covering of the erection chambers, known as "plaque". The appearance of indurated plaque and a resultant curvature or indentation is a well described medical condition known as "Peyronie's Disease" and may occur in men who did or did not undergo radical prostatectomy. The purpose of this study is to evaluate these changes in penile shape and dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 21 years or older (no maximum age limit)
* Ability and willingness to give informed consent
* Clinically localized prostate cancer
* Open, laparoscopic or robotic-assisted radical prostatectomy
* Must be sexually active (penetrative or non-penetrative sexual encounters, either with a partner or self-stimulation)

Exclusion Criteria:

* Preoperative / Postoperative pelvic radiation therapy
* Preoperative / Postoperative hormonal treatment
* Preoperative Peyronie's disease
* Preoperative presence of a penile implant

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open, laparoscopic, or robotic-assisted laparoscopic radical prostatectomy at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2008-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assess the impact of radical retropubic prostatectomy on penile dimensions. | conclusion of the study
Assess the impact of radical retropubic prostatectomy on the development of Peyronie's Disease. | conclusion of the study

SECONDARY OUTCOMES:
Assess the association between penile length change and erectile function. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: John Mulhall, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States